CLINICAL TRIAL: NCT00782834
Title: Evaluation of Nilotinib in Advanced GIST Previously Treated With Imatinib and Sunitinib
Brief Title: Nilotinib in Advanced Gastrointestinal Stromal Tumors (GIST)
Acronym: 07060
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped early for futility, unable to meet accrual goals
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107DUS05T
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST; Nilotinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nilotinib — 400 mg orally twice daily until disease progression, intolerability or withdrawal of consent
  Other Names: Tasigna

SUMMARY:
This is a phase II study of Nilotinib for patients with advanced GIST that cannot be surgically removed. Patients are candidates for the study if their tumors have progressed on imatinib and sunitinib or if they were intolerant to these drugs. Patients may have received other investigational therapies as well. We are testing the benefit of nilotinib in advanced GIST looking at the length of time disease is controlled as well as the response of the disease to the drug.

DETAILED DESCRIPTION:
Nilotinib is an oral drug. The dose is 400 mg twice daily

Patients are evaluated every 8 weeks for disease response. Blood work is assessed for safety initially weekly, then every 4 weeks. Physical exams are performed initially weekly and then decreased to every 4 weeks after the first month.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically or cytologically confirmed GIST
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 millimeters (mm) with conventional techniques or as >= 10 mm with spiral CT scan.
* Patients may have received prior chemotherapy or radiation therapy. Patients must have recovered from any prior therapy and at least 4 weeks (6 weeks for nitrosoureas or mitomycin C; 2 weeks for limited field palliative radiation) must have elapsed since prior treatment.
* Patients must have received and progressed on imatinib and sunitinib. Except for nilotinib, patients may have received additional tyrosine kinase inhibitors or additional targeted therapies.
* Age >= 18 years.
* Life expectancy of greater than 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count >= 1,500/mcL
  * platelets >= 100,000/mcL
  * total bilirubin <= 1.5 times Upper Limits of Normal (ULN)
  * AST(SGOT)/ALT(SGPT) <= 2.5 X ULN OR <= 5.0 X ULN if considered due to tumor
  * Potassium, magnesium normal or corrected to normal limits prior to initiating drug
  * Calcium, phosphorus normal or corrected to normal limits prior to initiating drug
  * creatinine within normal institutional limits
  * creatinine clearance 24 hour creatinine clearance >= 50 mL/min (calculation by cockroft formula is acceptable)
* The effects of Nilotinib on the developing human fetus at the recommended therapeutic dose are unknown. Men or women of childbearing potential (WOCBP), to include female partners of heterosexual or bisexual patients, must agree to use an effective method of contraception during the study and for up to three months following termination of the study. Post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patients may not be receiving any other investigational agents within 4 weeks.
* Prior or concomitant malignancies (with a relapse in the last 5 years or requiring active treatment) other than GIST and with the exception of previous or concomitant basal cell skin cancer, previous cervical carcinoma in situ
* Impaired cardiac function at baseline, including any one of the following:

  * Left Ventricular Ejection Fraction (LVEF)< 45% or below the institutional Lower Limits of Normal (LLN) range (whichever is higher)
  * Complete left bundle branch block
  * Use of a ventricular paced cardiac pacemaker
  * Congenital long QT syndrome or family history of long QT syndrome
  * History of or presence of significant ventricular or atrial tachyarrhythmias
  * Clinically significant resting bradycardia (< 50 beats per minute)
  * QTc > 450 msec on screening ECG (using the QTcF formula). If QTc > 450 msec and electrolytes are not within normal ranges (electrolytes should be corrected and then the patient rescreened for QTc.
  * Right bundle branch block plus left anterior hemiblock, bifascicular block
  * Myocardial infarction within 12 months prior to Visit 1
  * Other clinically significant heart disease (e.g., unstable angina, congestive heart failure or uncontrolled hypertension)
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol e.g. impairment of gastrointestinal (GI) function, or GI disease that may significantly alter the absorption of the study drugs, uncontrolled diabetes
* Use of therapeutic coumarin derivatives (i.e. warfarin, acenoucumarol, phenprocoumon)
* Use of any medications that prolong the QT interval and CYP3A4 inhibitors if the treatment cannot be either safely discontinued or switched to a different medication prior to starting study drug administration. Please see http://www.torsades.org/medical-pros/drug-lists/printable-drug-list.cfm for a comprehensive list of agents that prolong the QT interval as well as
* Patients who have undergone major surgery <= 2 weeks prior to Visit 1 or who have not recovered from side effects of such surgery
* A history of noncompliance to medical regimens or inability or unwillingness to return for scheduled visits, patients who are pregnant or breast feeding, and patients unwilling or unable to comply with the requirements for the protocol.
* Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-07; Primary Completion 2008-07 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were accrued between 7/03/2008 and 9/24/2009 at Fox Chase Cancer Center outpatient medical oncology clinics.
Pre-assignment Details: Advanced GIST with measurable disease; previously treated with at least imatinib and sunitinib; a 5-day washout from prior tyrosine kinase inhibitor therapy. Normal cardiac function with LVEF 45% or >, no history of significant heart disease,arrhythmias,congenital long QT sydrome, heart block, MI within 12 mos of visit 1 or unstable angina, CHF
Groups:
- Nilotinib Arm: All patients treated with nilotinib 400 mg BID orally daily; 4 weeks = one cycle
Period: Screened Patients
Arm/Group | Nilotinib Arm
Started | 15
Completed | 14 (1 pt ineligible d/t arrhythmia)
Not Completed | 1
Period: Treatment Phase
Arm/Group | Nilotinib Arm
Started | 14
Completed | 13
Not Completed | 1
Not completed — fibrous tumor not GIST | 1

BASELINE CHARACTERISTICS:
Population: Screened:
  Started: 15 patients Completed: 14 patients Comments: 1 patient deemed ineligible due to arrhythmia.
  Treatment Phase:
  Started: 14 patients Completed: 13 patients Comments: 1 patient on extensive pathology review was found to have a solitary fibrous tumor, not GIST.
Arm/Group | Nilotinib Arm
Number analyzed (Participants) | 15
Age Categorical [Number; unit: participants]
  <=18 years | 0 [0 to 18]
  Between 18 and 65 years | 9 [54 to 63]
  >=65 years | 4 [68 to 78]
Gender [Number; unit: participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 13
Primary Site of Cancer [Number; unit: Participants] — Stomach 6; Small bowel 5; Colon 1; Rectum 1
  Participants
    Stomach | 6
    Small Bowel | 5
    Colon | 1
    Rectum | 1
Prior Tyrosine Kinase Inhibitor (TKI) [Number; unit: Participants] — Imatinib (IM) + Sunitinib (SU); Imatinib + Sunitinib + Nasatinib (NA); Imatinib +Sunitinib + Radiotherapy (RT) + Chemotherapy (CT)
  Participants
    IM and SU | 11
    IM, SU and NA | 1
    IM, SU, RT and CT | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate at 6 Months
Description: Number of participants that demonstrate progression free survival at 6 months
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Nilotinib Arm
Number analyzed (Participants) | 13
Participants | 13

2. Primary Outcome: Response Rate
Description: Response rate of nilotinib by RECIST criteria evaluated every 2 months for the first 6 months then every 3 months for the duration of treatment period.
Time Frame: 1year
Measure: Number; unit: Participants
Arm/Group | Nilotinib Arm
Number analyzed (Participants) | 13
Participants | 5

ADVERSE EVENTS:
Arm/Group | Nilotinib Arm
Serious Adverse Events (participants affected / at risk) | 12/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nilotinib Arm (N=13)
Pain associated with constipation (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Nausea vomiting weakness followed by death (Gastrointestinal disorders) | 1 (1)
Profound weakness (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Severe abdominal pain (Gastrointestinal disorders) | 1 (1)
Severe anemia (Blood and lymphatic system disorders) | 1 (1)
Altered mental status dec pulse ox (Psychiatric disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Acute azotemia (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nilotinib Arm (N=13)
Leukopenia (Blood and lymphatic system disorders) | 6 (7)
Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 12 (23)
Urinary tract infection (Infections and infestations) | 1 (2)
Fatigue (General disorders) | 13 (23)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (9)
Edema (Cardiac disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 5 (9)
Vomiting (Gastrointestinal disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 7 (12)
Diarrhea (Gastrointestinal disorders) | 3 (7)
Constipation (Gastrointestinal disorders) | 7 (10)
GI Pain (Gastrointestinal disorders) | 5 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Creatinine (Investigations) | 4 (5)
Alk Phos (Investigations) | 6 (10)
SGOT (Investigations) | 4 (7)
Bilirubin (Investigations) | 2 (3)
Lipase (Investigations) | 2 (2)
Hypoalbuminemia (Investigations) | 6 (9)
Hyponatremia (Investigations) | 4 (6)
Hyperkalemia (Investigations) | 5 (8)
Hypocalcemia (Investigations) | 1 (1)
Hypomagnesemia (Investigations) | 4 (4)
Hoarseness voice changes (General disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (7)

LIMITATIONS AND CAVEATS:
The study failed to meet its accrual goals. Study terminated prior to accruing 17 subjects due to futility of meeting endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No